CLINICAL TRIAL: NCT03984019
Title: Cardiac Changes After Stereotactic Radiotherapy for Early Stage NSCLC Cancer or Lung Metastasis
Acronym: HALO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual due to COVID-19 and lower accrual than expected.
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: M19CCR
Record Dates: First submitted 2019-05-21; First posted 2019-06-12 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer Stage I; Lung Cancer Stage II; Lung Metastases
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an exploratory study to determine whether cardiac changes occur after radiation treatment. Patients are treated following standard clinical practice, with additional diagnostic investigations. The study design is therefore a cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A (Other): Radiotherapy; SBRT Additional cardiac diagnostics
  Interventions: Diagnostic Test: Cardiac condition measurements

INTERVENTIONS:
Diagnostic Test: Cardiac condition measurements — Cardiac MRI, ECG, echocardiography, cardiac blood markers

SUMMARY:
The investigators aim to optimize the radiation treatment of early stage lung cancer patients. Therefore, detailed understanding is needed of the type of toxicity and the location of these toxicities for patients who receive high fraction doses. These have not been measured in these patients before, therefore our primary research question is: is it possible to measure changes in cardiac condition after radiotherapy, with respect to cardiac arrhythmias, fibrosis, hemodynamic function change and pericarditis?

DETAILED DESCRIPTION:
Rationale: For lung cancer patients that receive thoracic irradiation, cardiac toxicity was not considered to play a role, because it was expected to occur many years after treatment. However, recently several studies have shown higher death rates for lung cancer patients receiving higher cardiac doses, possibly due to cardiac toxicity. Most knowledge on cardiac toxicity that is available, is based on patients that receive conventionally fractionated radiation treatment, where the heart receives a relatively low dose of radiation. For patients that receive stereotactic body radiation therapy (SBRT), which gives high fraction doses, the heart may receive peak doses of radiation, especially for centrally located lung tumours. This type of therapy is standard of care for early stage lung cancer patients, with very high local control that is similar to surgically treated patients. In order to improve the radiation treatment for these early stage lung cancer patients, detailed knowledge on cardiac toxicity in these patients is necessary.

Objective: the investigators aim to optimize the radiation treatment of early stage lung cancer patients. To reach that goal, detailed understanding is needed of the type of toxicity and the location on the heart of these toxicities for patients who receive high fraction doses. These have not been measured in this category of patients before, therefore our primary research question is: is it possible to measure changes in cardiac condition 3 or 12 months after radiotherapy, with respect to cardiac arrhythmias, tissue fibrosis, hemodynamic function change and pericarditis? Our secondary research question is: is it possible to measure local fibrosis and correlate this to local dose? The third research question is: is it possible to measure early cardiac morphology changes during the course of the irradiation? Study design: Twenty five patients with early stage lung cancer or a solitary lung metastasis of a solid tumour, who are treated with SBRT will be enrolled in an observational prospective cohort study and treated following standard clinical practice on a cone-beam or MR guided linear accelerator (Linac). Condition of the heart will be examined before treatment using ECG, cardiac MRI with added T1- and T2-mapping, echocardiography and blood biomarkers. These tests will be repeated 3 and 12 months after treatment.

Study population: 25 patients with a lung tumour in close proximity to the heart (edge of tumour <3cm from the heart) will be included. All patients receive SBRT for a primary lung tumour (stage IA-IIB), or for a solitary lung metastasis of a solid tumour.

Intervention (if applicable): not applicable Main study parameters/endpoints: It will be investigated 1) if changes in cardiac condition (cardiac arrhythmias, fibrosis, hemodynamic function change and pericarditis) can be visualised and quantified. A negative change of more than 5% between pre-and post-treatment measurements is considered toxicity. 2) If local fibrosis is associated to local dose, 3) if morphology changes are visible during treatment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The patient will have 3 sessions with several diagnostic tests: ECGs, cardiac MRIs, echocardiography and blood sampling, and will fill out 3 questionnaires. Limited side effects of these tests are expected. Cardiac tests will be evaluated by a cardiologist and dedicated radiologist and reported to the radiation oncologist who will inform the patient and refer to the cardiologist if needed. The burden for these patients will be, next to the time spent for the diagnostic tests and travel time; an intravenous blood sampling and administration of MRI contrast agent. The additional time spent for diagnostic tests per session are: echo (30 min), ECG (5 min), vena puncture (5 min) and MRI (45 min) + time in the waiting room. Filling out the 3 questionnaires will take 15 min each. The possible benefit for the patient is the extensive cardiac screening. Should a problem come to light, the patient will be referred to the cardiologist.

Results from this patient cohort are directly relatable to all early stage NSCLC who are treated with SBRT, and possibly oesophageal cancer patients as well. Should this study show that cardiac dose causes cardiac toxicity in this time frame, the aim should be to improve treatment for all patients who are comparable. Ergo, patients who receive cardiac dose because of their tumour location, and who are generally unfit for surgery because of their physical condition (early stage NSCLC patients and oesophageal cancer patients).

ELIGIBILITY:
Inclusion Criteria:

* Receive SBRT treatment for stage 1A-2B NSCLC or for a solitary lung metastasis of a solid tumour
* Closest distance between edge of tumor and heart < 3 cm

Exclusion Criteria:

* Pacemaker/ICD
* Renal function below GFR <30 ml/min/1.7m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a change in cardiac condition | 1 year
  Percentage of patients with at least 5% change in cardiac arrhythmia (outcome 2) and/or at least 5% change in fibrosis (outcome 3) and/or at least 5% change in hemodynamic function (outcome 4) and/or development of pericarditis post-treatment (outcome 5)
Percentage of change in cardiac arrhythmia | 1 year
  Percentage of change in ECG-derived QRS duration (s) between Pre- and Post-treatment values
Percentage of change in fibrosis | 1 year
  Percentage of change in MRI-derived Extra Cellular Volume (cc) between Pre- and Post-treatment values
Percentage of change in hemodynamic function | 1 year
  Percentage of change in MRI- and echocardiography-derived ejection fraction (%) between Pre- and Post-treatment values
Binary change in pericarditis status | 1 year
  Presence of pericarditis signs on MRI post-treatment while absence of pericarditis signs pre-treatment: yes/no

SECONDARY OUTCOMES:
Local fibrosis | 1 year
  Is there a correlation between the presence of local fibrosis and dose to this region
Morphology changes | 1 year
  Are changes in morphology visible on the MRI scans made during treatment, compared to the pre treatment MRIs

CONTACTS AND LOCATIONS:
Overall Officials: Jose Belderbos, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (3):
- Netherlands (3):
  - Netherlands Cancer Institute, Amsterdam
  - Amsterdam UMC, location AMC, Amsterdam
  - Leids Universitair Medisch Centrum (LUMC), Leiden

IPD SHARING:
Plan to Share IPD: No
No data will be shared